## Sustainable Football: Physical Profile, Training Load, Risk Factors and Injuries in Swedish Elite Football

Date: 2024-08-31

## Sustainable football: Physical profile, training load, risk factors and injuries in Swedish elite football

## Informed consent and consent regarding data processing in the study

| have had the opportunity to ask questi | he study and have read the above written information. I ons and have them answered. I am aware that my y voluntary and that I can cancel my participation at any |
|---|---|
| Name of the participant | |
| Participant's signature | Place and date |
| and your results will be processe them. During the data processing cannot be distinguished. Only the | stored in a register and processed. Your answers of so that unauthorized persons cannot access g, your data will be coded, so that an individual e person responsible for the study has access to study may be published, individual individuals |
| I agree that coded data about my electronically | person may be stored and processed |
| Name of the participant | |
| Participant's signature | Place and date |